CLINICAL TRIAL: NCT02596815
Title: Hypoalgesic Effect of Median Nerve Neural Mobilization in Cervicobrachial Pain Compared to a Controlled Group
Brief Title: Hypoalgesic Effect of Median Nerve Neural Mobilization Compared to a Controlled Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Francisco Unda Solano, PHD Student, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE0072015-3
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Cervicobrachial Neuralgia
MeSH Terms: conditions — Brachial Plexus Neuritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Median Nerve Neural Mobilization (Experimental): 15 minute Median Nerve Neural Mobilization sessions 3 times a week during 6 continuous weeks.The maximum degree of elbow extension applied in the Median Nerve neural mobilization procedure was determined through the use of a Universal Goniometer Device.
  Interventions: Procedure: Median Nerve Neural Mobilization; Device: Goniometer
- Waiting list control group (Active Comparator): Patients assigned to a 6 week waiting list to receive treatment
  Interventions: Procedure: Median Nerve Neural Mobilization; Device: Goniometer

INTERVENTIONS:
Procedure: Median Nerve Neural Mobilization — Nonsurgical noninvasive Median Nerve neural mobilization procedure was applied by a physical therapist continuously during 2 minutes in 5 different occasions with 1 minute of rest between each 2 minute application of the Neural Mobilization technique. The intervention was applied during a period of 6 weeks. The maximum level of elbow extension movement degree without the reproduction of symptoms during the application of the Median Nerve Neural mobilization treatment was determined through the baseline use of a Universal Goniometer Device.
  Other Names: Neural Tissue Mobilization of the Median Nerve; Median Nerve Neurodynamics
Device: Goniometer

SUMMARY:
The purpose of these study is to compare the effectivity of the Median Nerve Neural Mobilization technique to the complete absence of treatment in a group of patients who suffer cervicobrachial pain.

DETAILED DESCRIPTION:
Median Nerve Neural Mobilization (MNNM) is a non invasive physical therapy technique that achieves pain relief through mechanical stimulation of the Median Nerve and the brachial plexus. It is believed that the hypoalgesic effect offered by the neural tissue mobilization procedure is a consequence of descending nervous system pain modulation activity and an improvement in the distinct biomechanical and sensitive properties of the involved neural tissue. The neural tissue mobilization procedure is associated to an increase in nerve mobility, edema, inflammation and intraneural pressure reduction without any known side effects when applied properly which is an important contrast to the wide variety of side effects caused by commonly used drug therapy to treat cervicobrachial pain.

Despite the crescent interest among the scientific community in evidence based options to treat pain there is a current lack of enough controlled double blind clinical trials that measure the effectiveness of neural tissue mobilization techniques such as the (MNNM) and its specific effect over cervicobrachial pain. For this reason the present investigation consisted in the application of a treatment protocol based on Median Nerve Neural Mobilization in a controlled double blind clinical trial with the aim to assess its clinical effectiveness in treating pain symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cervicobrachial pain confirmed by magnetic resonance imaging
* Presence of unilateral symptoms of arm pain, paresthesia or numbness in the upper extremity during at least 3 continuous months previous to the application of treatment.
* Positive results in all of the following tests: Spurling, Distraction, and Upper Limb

Exclusion Criteria:

* Contraindication in the use of nonsteroidal anti-inflammatory drugs (NSAIDs)
* The use of any type of treatment, therapy, procedure or drug to relieve pain
* Patients who are under anticonvulsant, antidepressant or psychotropic medication
* Vertebral instability
* Vertebral osteoporosis
* Vertebral or spine infection.
* Neurologic diseases of genetic, infectious or neoplastic origin
* Cervical stenosis myelopathy
* Pregnancy
* Kinesiophobia
* Endocrine disorders and menopause
* History of spine surgery
* Intellectual disability, severe mental illness, intoxication, severe sleep deprivation, Alzheimer's disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline using the Numeric Rating Scale for Pain at 1 hour | at baseline for both arms and 1 hour after the application of treatment only in the experimental arm, corresponding to intervention days 1, 9 and 18.
  the Numeric Rating scale for Pain (NRS) is an 11 point scale for patient self reporting of pain in which 0 points represents the total absence of pain and 10 points the worst state of pain, it was employed to evaluate the presence and relieve of cervicobrachial pain symptoms.

SECONDARY OUTCOMES:
Change from baseline of the Physical function involving the affected upper limb using the Quik DASH Scale | at baseline, corresponding to intervention days 1 and 18 of treatment
  The disabilities of the arm quick test (Quick DASH) is a self report short questionnaire designed to measure physical function and symptoms in people with any or several musculoskeletal disorders of the upper limb.
Cervical Rotation Range of Motion (CROM) | at baseline for both arms and 1 hour after the application of treatment only in the experimental arm, corresponding to intervention days 1 and 18 .
  Cervical rotation was assessed in units of rotation degrees, using the cervical range of motion device (CROM).

CONTACTS AND LOCATIONS:
Overall Officials: Francisco H Unda, PT, MSc, Principal Investigator — Universidad Europea de Madrid
Locations (2):
- Venezuela (2):
  - Centro Médico y de Especialidades Pediátricas Dr. José Gregorio Hernández, San Diego, Carabobo
  - Centro de Medicina Fisica y de Rehabilitacion FISIOREH, Valencia, Carabobo

REFERENCES:
- [Background] Turajane T, Wongbunnak R, Patcharatrakul T, Ratansumawong K, Poigampetch Y, Songpatanasilp T. Gastrointestinal and cardiovascular risk of non-selective NSAIDs and COX-2 inhibitors in elderly patients with knee osteoarthritis. J Med Assoc Thai. 2009 Dec;92 Suppl 6:S19-26. PMID 20128070
- [Result] Cowell IM, Phillips DR. Effectiveness of manipulative physiotherapy for the treatment of a neurogenic cervicobrachial pain syndrome: a single case study -- experimental design. Man Ther. 2002 Feb;7(1):31-8. doi: 10.1054/math.2001.0429. PMID 11884154
- [Result] Salt E, Wright C, Kelly S, Dean A. A systematic literature review on the effectiveness of non-invasive therapy for cervicobrachial pain. Man Ther. 2011 Feb;16(1):53-65. doi: 10.1016/j.math.2010.09.005. Epub 2010 Nov 12. PMID 21075037
- [Result] Allison GT, Nagy BM, Hall T. A randomized clinical trial of manual therapy for cervico-brachial pain syndrome -- a pilot study. Man Ther. 2002 May;7(2):95-102. doi: 10.1054/math.2002.0453. PMID 12151246
- [Result] Huisstede BM, Bierma-Zeinstra SM, Koes BW, Verhaar JA. Incidence and prevalence of upper-extremity musculoskeletal disorders. A systematic appraisal of the literature. BMC Musculoskelet Disord. 2006 Jan 31;7:7. doi: 10.1186/1471-2474-7-7. PMID 16448572
- [Result] Radhakrishnan K, Litchy WJ, O'Fallon WM, Kurland LT. Epidemiology of cervical radiculopathy. A population-based study from Rochester, Minnesota, 1976 through 1990. Brain. 1994 Apr;117 ( Pt 2):325-35. doi: 10.1093/brain/117.2.325. PMID 8186959
- [Result] Daffner SD, Hilibrand AS, Hanscom BS, Brislin BT, Vaccaro AR, Albert TJ. Impact of neck and arm pain on overall health status. Spine (Phila Pa 1976). 2003 Sep 1;28(17):2030-5. doi: 10.1097/01.BRS.0000083325.27357.39. PMID 12973155
- [Result] Isabel de-la-Llave-Rincon A, Puentedura EJ, Fernandez-de-Las-Penas C. Clinical presentation and manual therapy for upper quadrant musculoskeletal conditions. J Man Manip Ther. 2011 Nov;19(4):201-11. doi: 10.1179/106698111X13129729551985. PMID 23115473
- [Result] Antonelli BA, de Paula Xavier AA, Oenning P, Baumer MH, da Silva TF, Pilatti LA. Prevalence of cervicobrachial discomforts in elementary school teachers. Work. 2012;41 Suppl 1:5709-14. doi: 10.3233/WOR-2012-0927-5709. PMID 22317661
- [Result] Dillingham TR. Evaluating the patient with suspected radiculopathy. PM R. 2013 May;5(5 Suppl):S41-9. doi: 10.1016/j.pmrj.2013.03.015. Epub 2013 Mar 19. PMID 23524070
- [Result] Boyles R, Toy P, Mellon J Jr, Hayes M, Hammer B. Effectiveness of manual physical therapy in the treatment of cervical radiculopathy: a systematic review. J Man Manip Ther. 2011 Aug;19(3):135-42. doi: 10.1179/2042618611Y.0000000011. PMID 22851876
- [Result] Eubanks JD. Cervical radiculopathy: nonoperative management of neck pain and radicular symptoms. Am Fam Physician. 2010 Jan 1;81(1):33-40. PMID 20052961
- [Result] Peolsson A, Soderlund A, Engquist M, Lind B, Lofgren H, Vavruch L, Holtz A, Winstrom-Christersson A, Isaksson I, Oberg B. Physical function outcome in cervical radiculopathy patients after physiotherapy alone compared with anterior surgery followed by physiotherapy: a prospective randomized study with a 2-year follow-up. Spine (Phila Pa 1976). 2013 Feb 15;38(4):300-7. doi: 10.1097/BRS.0b013e31826d2cbb. PMID 23407407
- [Result] Caridi JM, Pumberger M, Hughes AP. Cervical radiculopathy: a review. HSS J. 2011 Oct;7(3):265-72. doi: 10.1007/s11420-011-9218-z. Epub 2011 Sep 9. PMID 23024624
- [Result] Young IA, Michener LA, Cleland JA, Aguilera AJ, Snyder AR. Manual therapy, exercise, and traction for patients with cervical radiculopathy: a randomized clinical trial. Phys Ther. 2009 Jul;89(7):632-42. doi: 10.2522/ptj.20080283. Epub 2009 May 21. PMID 19465371
- [Result] Campbell WW. Evaluation and management of peripheral nerve injury. Clin Neurophysiol. 2008 Sep;119(9):1951-65. doi: 10.1016/j.clinph.2008.03.018. Epub 2008 May 14. PMID 18482862
- [Result] Walton Walter WJ. Brain´s Diseases Of The Nervous System. London: Oxford UP; 1969
- [Result] Nikolaidis I, Fouyas IP, Sandercock PA, Statham PF. Surgery for cervical radiculopathy or myelopathy. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD001466. doi: 10.1002/14651858.CD001466.pub3. PMID 20091520
- [Result] Legakis A, Boyd BS. The influence of scapular depression on upper limb neurodynamic test responses. J Man Manip Ther. 2012 May;20(2):75-82. doi: 10.1179/2042618611Y.0000000020. PMID 23633886
- [Result] McGregor AH, Probyn K, Cro S, Dore CJ, Burton AK, Balague F, Pincus T, Fairbank J. Rehabilitation following surgery for lumbar spinal stenosis. Cochrane Database Syst Rev. 2013 Dec 9;2013(12):CD009644. doi: 10.1002/14651858.CD009644.pub2. PMID 24323844
- [Result] Cleland JA, Whitman JM, Fritz JM, Palmer JA. Manual physical therapy, cervical traction, and strengthening exercises in patients with cervical radiculopathy: a case series. J Orthop Sports Phys Ther. 2005 Dec;35(12):802-11. doi: 10.2519/jospt.2005.35.12.802. PMID 16848101
- [Result] Beneciuk JM, Bishop MD, George SZ. Effects of upper extremity neural mobilization on thermal pain sensitivity: a sham-controlled study in asymptomatic participants. J Orthop Sports Phys Ther. 2009 Jun;39(6):428-38. doi: 10.2519/jospt.2009.2954. PMID 19487826
- [Result] Elvey R HT. Neural tissue evaluation and treatment, Donatelli R, Physical Therapy of the Shoulder,. 3rd ed. Livingstone C, editor. New York; 1997
- [Result] Fritz JM, Thackeray A, Brennan GP, Childs JD. Exercise only, exercise with mechanical traction, or exercise with over-door traction for patients with cervical radiculopathy, with or without consideration of status on a previously described subgrouping rule: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Feb;44(2):45-57. doi: 10.2519/jospt.2014.5065. Epub 2014 Jan 9. PMID 24405257
- [Result] Persson LC, Carlsson CA, Carlsson JY. Long-lasting cervical radicular pain managed with surgery, physiotherapy, or a cervical collar. A prospective, randomized study. Spine (Phila Pa 1976). 1997 Apr 1;22(7):751-8. doi: 10.1097/00007632-199704010-00007. PMID 9106315
- [Result] Carlesso LC, Macdermid JC, Gross AR, Walton DM, Santaguida PL. Treatment preferences amongst physical therapists and chiropractors for the management of neck pain: results of an international survey. Chiropr Man Therap. 2014 Mar 24;22(1):11. doi: 10.1186/2045-709X-22-11. PMID 24661461
- [Result] Coppieters MW, Stappaerts KH, Wouters LL, Janssens K. The immediate effects of a cervical lateral glide treatment technique in patients with neurogenic cervicobrachial pain. J Orthop Sports Phys Ther. 2003 Jul;33(7):369-78. doi: 10.2519/jospt.2003.33.7.369. PMID 12918862
- [Result] Garland EL. Treating chronic pain: the need for non-opioid options. Expert Rev Clin Pharmacol. 2014 Sep;7(5):545-50. doi: 10.1586/17512433.2014.928587. Epub 2014 Jun 11. PMID 24918159
- [Result] Santos FM, Grecco LH, Pereira MG, Oliveira ME, Rocha PA, Silva JT, Martins DO, Miyabara EH, Chacur M. The neural mobilization technique modulates the expression of endogenous opioids in the periaqueductal gray and improves muscle strength and mobility in rats with neuropathic pain. Behav Brain Funct. 2014 May 13;10:19. doi: 10.1186/1744-9081-10-19. PMID 24884961
- [Result] Ogneva IV. Cell mechanosensitivity: mechanical properties and interaction with gravitational field. Biomed Res Int. 2013;2013:598461. doi: 10.1155/2013/598461. Epub 2012 Dec 26. PMID 23509748
- [Result] Bonin RP, Bories C, De Koninck Y. A simplified up-down method (SUDO) for measuring mechanical nociception in rodents using von Frey filaments. Mol Pain. 2014 Apr 16;10:26. doi: 10.1186/1744-8069-10-26. PMID 24739328
- [Result] Moriarty O, Finn DP. Cognition and pain. Curr Opin Support Palliat Care. 2014 Jun;8(2):130-6. doi: 10.1097/SPC.0000000000000054. PMID 24722475
- [Result] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Result] Courtney CA, Clark JD, Duncombe AM, O'Hearn MA. Clinical presentation and manual therapy for lower quadrant musculoskeletal conditions. J Man Manip Ther. 2011 Nov;19(4):212-22. doi: 10.1179/106698111X13129729552029. PMID 23115474
- [Result] Woolf CJ, Salter MW. Neuronal plasticity: increasing the gain in pain. Science. 2000 Jun 9;288(5472):1765-9. doi: 10.1126/science.288.5472.1765. PMID 10846153
- [Result] Woolf CJ. Central sensitization: uncovering the relation between pain and plasticity. Anesthesiology. 2007 Apr;106(4):864-7. doi: 10.1097/01.anes.0000264769.87038.55. No abstract available. PMID 17413924
- [Result] Santos FM, Silva JT, Giardini AC, Rocha PA, Achermann AP, Alves AS, Britto LR, Chacur M. Neural mobilization reverses behavioral and cellular changes that characterize neuropathic pain in rats. Mol Pain. 2012 Jul 29;8:57. doi: 10.1186/1744-8069-8-57. PMID 22839415
- [Result] Villafane JH. Botulinum toxin type A combined with neurodynamic mobilization for lower limb spasticity: a case report. J Chiropr Med. 2013 Mar;12(1):39-44. doi: 10.1016/j.jcm.2013.01.001. PMID 23997723
- [Result] Villafane JH, Pillastrini P, Borboni A. Manual therapy and neurodynamic mobilization in a patient with peroneal nerve paralysis: a case report. J Chiropr Med. 2013 Sep;12(3):176-81. doi: 10.1016/j.jcm.2013.10.007. PMID 24396318
- [Result] Ellis RF, Hing WA, McNair PJ. Comparison of longitudinal sciatic nerve movement with different mobilization exercises: an in vivo study utilizing ultrasound imaging. J Orthop Sports Phys Ther. 2012 Aug;42(8):667-75. doi: 10.2519/jospt.2012.3854. Epub 2012 Jun 18. PMID 22711174
- [Result] Shacklock M. Neural mobilization: a systematic review of randomized controlled trials with an analysis of therapeutic efficacy. J Man Manip Ther. 2008;16(1):23-4. doi: 10.1179/106698108790818602. No abstract available. PMID 19119381
- [Result] Lin PL, Shih YF, Chen WY, Ma HL. Neurodynamic responses to the femoral slump test in patients with anterior knee pain syndrome. J Orthop Sports Phys Ther. 2014 May;44(5):350-7. doi: 10.2519/jospt.2014.4781. Epub 2014 Apr 14. PMID 24730437
- [Result] Franze K. The mechanical control of nervous system development. Development. 2013 Aug;140(15):3069-77. doi: 10.1242/dev.079145. PMID 23861056
- [Result] Livne A, Bouchbinder E, Geiger B. Cell reorientation under cyclic stretching. Nat Commun. 2014 May 30;5:3938. doi: 10.1038/ncomms4938. PMID 24875391
- [Result] Lopez-Fagundo C, Bar-Kochba E, Livi LL, Hoffman-Kim D, Franck C. Three-dimensional traction forces of Schwann cells on compliant substrates. J R Soc Interface. 2014 Aug 6;11(97):20140247. doi: 10.1098/rsif.2014.0247. PMID 24872498
- [Result] Nee RJ, Vicenzino B, Jull GA, Cleland JA, Coppieters MW. Neural tissue management provides immediate clinically relevant benefits without harmful effects for patients with nerve-related neck and arm pain: a randomised trial. J Physiother. 2012;58(1):23-31. doi: 10.1016/S1836-9553(12)70069-3. PMID 22341379
- [Result] Savva C, Giakas G. The effect of cervical traction combined with neural mobilization on pain and disability in cervical radiculopathy. A case report. Man Ther. 2013 Oct;18(5):443-6. doi: 10.1016/j.math.2012.06.012. Epub 2012 Jul 18. PMID 22818658
- [Result] Ellis RF, Hing WA. Neural mobilization: a systematic review of randomized controlled trials with an analysis of therapeutic efficacy. J Man Manip Ther. 2008;16(1):8-22. doi: 10.1179/106698108790818594. PMID 19119380
- [Result] Cueco T. La columna cervical ; Sindromes clínicos y su tratamiento manipulativo. Panamericano E, editor. 2008. 40-41 p.
- [Result] Hsu E, Argof C, Galluzi K DA. Problem based pain management. Press CU, editor. 2013. 57 p.
- [Result] Basson A, Olivier B, Ellis R, Coppieters M, Stewart A, Mudzi W. The effectiveness of neural mobilizations in the treatment of musculoskeletal conditions: a systematic review protocol. JBI Database System Rev Implement Rep. 2015 Jan;13(1):65-75. doi: 10.11124/jbisrir-2015-1401. PMID 26447008
- [Result] Niemisto L, Kalso E, Malmivaara A, Seitsalo S, Hurri H. Radiofrequency denervation for neck and back pain. A systematic review of randomized controlled trials. Cochrane Database Syst Rev. 2003;(1):CD004058. doi: 10.1002/14651858.CD004058. PMID 12535508
- [Result] van Tulder M, Malmivaara A, Koes B. Repetitive strain injury. Lancet. 2007 May 26;369(9575):1815-1822. doi: 10.1016/S0140-6736(07)60820-4. PMID 17531890
- [Result] Mico JA, Ardid D, Berrocoso E, Eschalier A. Antidepressants and pain. Trends Pharmacol Sci. 2006 Jul;27(7):348-54. doi: 10.1016/j.tips.2006.05.004. Epub 2006 Jun 9. PMID 16762426
- [Result] Carson VB. Mental health nursing: the nurse-patient journey W.B. Saunders. 2000: p. 423
- [Result] van der Velde G, Hogg-Johnson S, Bayoumi AM, Cassidy JD, Cote P, Boyle E, Llewellyn-Thomas H, Chan S, Subrata P, Hoving JL, Hurwitz E, Bombardier C, Krahn M. Identifying the best treatment among common nonsurgical neck pain treatments: a decision analysis. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S209-18. doi: 10.1016/j.jmpt.2008.11.021. PMID 19251067
- [Result] Sella G. Practical Guide to Chronic Pain Syndromes Compression Neuropathies Chap 8. Press C, editor. 2009. 85-98 p.
- [Result] Borenstein D. Low Back and Neck Pain. Low Back and Neck Pain [Internet]. 2004. p. 771-849. Available from: http://www.sciencedirect.com/science/ article/pii/B9780721692777500283
- [Result] Sniezek PJ, Brodland DG, Zitelli JA. A randomized controlled trial comparing acetaminophen, acetaminophen and ibuprofen, and acetaminophen and codeine for postoperative pain relief after Mohs surgery and cutaneous reconstruction. Dermatol Surg. 2011 Jul;37(7):1007-13. doi: 10.1111/j.1524-4725.2011.02022.x. Epub 2011 May 11. PMID 21561527
- [Result] Jeyakumar A, Brickman TM, Williamson ME, Hirose K, Krakovitz P, Whittemore K, Discolo C. Nonsteroidal anti-inflammatory drugs and postoperative bleeding following adenotonsillectomy in pediatric patients. Arch Otolaryngol Head Neck Surg. 2008 Jan;134(1):24-7. doi: 10.1001/archoto.2007.11. PMID 18209131
- [Result] Kanabar D. A practical approach to the treatment of low-risk childhood fever. Drugs R D. 2014 Jun;14(2):45-55. doi: 10.1007/s40268-014-0052-x. PMID 24916274
- [Result] Moore RA, Derry S, Wiffen PJ, Straube S, Aldington DJ. Overview review: Comparative efficacy of oral ibuprofen and paracetamol (acetaminophen) across acute and chronic pain conditions. Eur J Pain. 2015 Oct;19(9):1213-23. doi: 10.1002/ejp.649. Epub 2014 Dec 22. PMID 25530283
- [Result] Kissin I. Scientometric assessment of drugs for chronic pain, 1979-2013: rapid growth of publications, paucity of successful drugs. J Pain Res. 2014 Aug 20;7:505-14. doi: 10.2147/JPR.S67479. eCollection 2014. PMID 25187736
- [Result] Nasca RJ. Cervical radiculopathy: current diagnostic and treatment options. J Surg Orthop Adv. 2009 Spring;18(1):13-8. PMID 19327260
- [Result] Fountas KN, Kapsalaki EZ, Nikolakakos LG, Smisson HF, Johnston KW, Grigorian AA, Lee GP, Robinson JS Jr. Anterior cervical discectomy and fusion associated complications. Spine (Phila Pa 1976). 2007 Oct 1;32(21):2310-7. doi: 10.1097/BRS.0b013e318154c57e. PMID 17906571
- [Result] Ghobrial GM, Viereck MJ, Margiotta PJ, Beygi S, Maulucci CM, Heller JE, Vaccaro AR, Harrop JS. Surgical management in 40 consecutive patients with cervical spinal epidural abscesses: shifting toward circumferential treatment. Spine (Phila Pa 1976). 2015 Sep 1;40(17):E949-53. doi: 10.1097/BRS.0000000000000942. PMID 25893350
- [Result] Persson LC, Moritz U, Brandt L, Carlsson CA. Cervical radiculopathy: pain, muscle weakness and sensory loss in patients with cervical radiculopathy treated with surgery, physiotherapy or cervical collar. A prospective, controlled study. Eur Spine J. 1997;6(4):256-66. doi: 10.1007/BF01322448. PMID 9294750
- [Result] Imani F, Motavaf M, Safari S, Alavian SM. The therapeutic use of analgesics in patients with liver cirrhosis: a literature review and evidence-based recommendations. Hepat Mon. 2014 Oct 11;14(10):e23539. doi: 10.5812/hepatmon.23539. eCollection 2014 Oct. PMID 25477978
- [Result] Asghar W, Jamali F. The effect of COX-2-selective meloxicam on the myocardial, vascular and renal risks: a systematic review. Inflammopharmacology. 2015 Feb;23(1):1-16. doi: 10.1007/s10787-014-0225-9. Epub 2014 Dec 17. PMID 25515365
- [Result] Unzueta A, Vargas HE. Nonsteroidal anti-inflammatory drug-induced hepatoxicity. Clin Liver Dis. 2013 Nov;17(4):643-56, ix. doi: 10.1016/j.cld.2013.07.009. Epub 2013 Sep 4. PMID 24099022
- [Result] Herndon CM, Dankenbring DM. Patient perception and knowledge of acetaminophen in a large family medicine service. J Pain Palliat Care Pharmacother. 2014 Jun;28(2):109-16. doi: 10.3109/15360288.2014.908993. Epub 2014 May 12. PMID 24813653
- [Result] Zadrazil J. [Nonsteroidal antiinflammatory drugs and the kidney]. Vnitr Lek. 2006 Jul-Aug;52(7-8):686-90. Czech. PMID 16967609
- [Result] Waddington F, Naunton M, Thomas J. Paracetamol and analgesic nephropathy: Are you kidneying me? Int Med Case Rep J. 2014 Dec 15;8:1-5. doi: 10.2147/IMCRJ.S71471. eCollection 2015. PMID 25548527
- [Result] Whelton A, Hamilton CW. Nonsteroidal anti-inflammatory drugs: effects on kidney function. J Clin Pharmacol. 1991 Jul;31(7):588-98. doi: 10.1002/j.1552-4604.1991.tb03743.x. PMID 1894754
- [Result] van der Linden MW, van der Bij S, Welsing P, Kuipers EJ, Herings RM. The balance between severe cardiovascular and gastrointestinal events among users of selective and non-selective non-steroidal anti-inflammatory drugs. Ann Rheum Dis. 2009 May;68(5):668-73. doi: 10.1136/ard.2007.087254. Epub 2008 May 21. PMID 18495734
- [Result] Ingrasciotta Y, Sultana J, Giorgianni F, Caputi AP, Arcoraci V, Tari DU, Linguiti C, Perrotta M, Nucita A, Pellegrini F, Fontana A, Cavagna L, Santoro D, Trifiro G. The burden of nephrotoxic drug prescriptions in patients with chronic kidney disease: a retrospective population-based study in Southern Italy. PLoS One. 2014 Feb 18;9(2):e89072. doi: 10.1371/journal.pone.0089072. eCollection 2014. PMID 24558471
- [Result] Pfizer Inc. Neurontin ® ( gabapentin ) Capsules Neurontin ® ( gabapentin ) Tablets Neurontin ® ( gabapentin ) Oral Solution. Neurontin Packag Inser. 2009;(LAB-01069.1):1-29.
- [Result] Aronson JK. Side Effects of Drugs Annual: A World Wide Yearly Survey of New Data in Adverse Drug Reactions. Newnes. 2014. p.1056-137
- [Result] Rodriguez SC, Olguin AM, Miralles CP, Viladrich PF. Characteristics of meningitis caused by Ibuprofen: report of 2 cases with recurrent episodes and review of the literature. Medicine (Baltimore). 2006 Jul;85(4):214-220. doi: 10.1097/01.md.0000229757.78057.50. PMID 16862046
- [Result] Auriel E, Regev K, Korczyn AD. Nonsteroidal anti-inflammatory drugs exposure and the central nervous system. Handb Clin Neurol. 2014;119:577-84. doi: 10.1016/B978-0-7020-4086-3.00038-2. PMID 24365321
- [Result] Bancos S, Bernard MP, Topham DJ, Phipps RP. Ibuprofen and other widely used non-steroidal anti-inflammatory drugs inhibit antibody production in human cells. Cell Immunol. 2009;258(1):18-28. doi: 10.1016/j.cellimm.2009.03.007. Epub 2009 Apr 5. PMID 19345936
- [Result] Volans G, Monaghan J, Colbridge M. Ibuprofen overdose. Int J Clin Pract Suppl. 2003 Apr;(135):54-60. PMID 12723749
- [Result] Moriarty O, McGuire BE, Finn DP. The effect of pain on cognitive function: a review of clinical and preclinical research. Prog Neurobiol. 2011 Mar;93(3):385-404. doi: 10.1016/j.pneurobio.2011.01.002. Epub 2011 Jan 7. PMID 21216272
- [Result] Krenkel O, Mossanen JC, Tacke F. Immune mechanisms in acetaminophen-induced acute liver failure. Hepatobiliary Surg Nutr. 2014 Dec;3(6):331-43. doi: 10.3978/j.issn.2304-3881.2014.11.01. PMID 25568858
- [Result] Jann MW, Slade JH. Antidepressant agents for the treatment of chronic pain and depression. Pharmacotherapy. 2007 Nov;27(11):1571-87. doi: 10.1592/phco.27.11.1571. PMID 17963465
- [Result] Salerno SM, Browning R, Jackson JL. The effect of antidepressant treatment on chronic back pain: a meta-analysis. Arch Intern Med. 2002 Jan 14;162(1):19-24. doi: 10.1001/archinte.162.1.19. PMID 11784215
- [Result] Fragemann K, Wiese C. Pain education policies and initiatives in Europe. J Pain Palliat Care Pharmacother. 2014 Dec;28(4):402-3. doi: 10.3109/15360288.2014.972004. Epub 2014 Oct 28. PMID 25348223
- [Result] Schug SA, Goddard C. Recent advances in the pharmacological management of acute and chronic pain. Ann Palliat Med. 2014 Oct;3(4):263-75. doi: 10.3978/j.issn.2224-5820.2014.10.02. PMID 25841906
- [Result] Wagner JG, Albert KS, Szpunar GJ, Lockwood GF. Pharmacokinetics of ibuprofen in man IV: absorption and disposition. J Pharmacokinet Biopharm. 1984 Aug;12(4):381-99. doi: 10.1007/BF01062664. PMID 6527231
- [Result] Rasu RS, Vouthy K, Crowl AN, Stegeman AE, Fikru B, Bawa WA, Knell ME. Cost of pain medication to treat adult patients with nonmalignant chronic pain in the United States. J Manag Care Spec Pharm. 2014 Sep;20(9):921-8. doi: 10.18553/jmcp.2014.20.9.921. PMID 25166291
- [Result] Chaparro LE, Wiffen PJ, Moore RA, Gilron I. Combination pharmacotherapy for the treatment of neuropathic pain in adults. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD008943. doi: 10.1002/14651858.CD008943.pub2. PMID 22786518
- [Result] Cohen SP, Hayek S, Semenov Y, Pasquina PF, White RL, Veizi E, Huang JH, Kurihara C, Zhao Z, Guthmiller KB, Griffith SR, Verdun AV, Giampetro DM, Vorobeychik Y. Epidural steroid injections, conservative treatment, or combination treatment for cervical radicular pain: a multicenter, randomized, comparative-effectiveness study. Anesthesiology. 2014 Nov;121(5):1045-55. doi: 10.1097/ALN.0000000000000409. PMID 25335172
- [Result] Schmid A, Brunner F, Wright A, Bachmann LM. Paradigm shift in manual therapy? Evidence for a central nervous system component in the response to passive cervical joint mobilisation. Man Ther. 2008 Oct;13(5):387-96. doi: 10.1016/j.math.2007.12.007. Epub 2008 Mar 3. PMID 18316238
- [Result] Harvey MP, Descarreaux M. Short term modulation of trunk neuromuscular responses following spinal manipulation: a control group study. BMC Musculoskelet Disord. 2013 Mar 13;14:92. doi: 10.1186/1471-2474-14-92. PMID 23496876
- [Result] McReynolds TM, Sheridan BJ. Intramuscular ketorolac versus osteopathic manipulative treatment in the management of acute neck pain in the emergency department: a randomized clinical trial. J Am Osteopath Assoc. 2005 Feb;105(2):57-68. PMID 15784928
- [Result] Dabbs V, Lauretti WJ. A risk assessment of cervical manipulation vs. NSAIDs for the treatment of neck pain. J Manipulative Physiol Ther. 1995 Oct;18(8):530-6. PMID 8583176
- [Result] Sheather-Reid RB, Cohen M. Efficacy of analgesics in chronic pain: a series of N-of-1 studies. J Pain Symptom Manage. 1998 Apr;15(4):244-52. doi: 10.1016/s0885-3924(98)00369-8. PMID 9601160
- [Result] Rainsford KD. Ibuprofen: from invention to an OTC therapeutic mainstay. Int J Clin Pract Suppl. 2013 Jan;(178):9-20. doi: 10.1111/ijcp.12055. PMID 23163543
- [Result] Vicenzino B, Collins D, Benson H, Wright A. An investigation of the interrelationship between manipulative therapy-induced hypoalgesia and sympathoexcitation. J Manipulative Physiol Ther. 1998 Sep;21(7):448-53. PMID 9777544
- [Result] X. Casado-Zumeta. Efectividad de la fisioterapia manual en el dolor cervicobraquial neuropático: una revisión sistematica. Fisioterapia. 2015;37(4).
- [Result] Brochwicz P, von Piekartz H, Zalpour C. Sonography assessment of the median nerve during cervical lateral glide and lateral flexion. Is there a difference in neurodynamics of asymptomatic people? Man Ther. 2013 Jun;18(3):216-9. doi: 10.1016/j.math.2012.10.001. Epub 2013 Jan 11. PMID 23317635
- [Result] Wang WT, Olson SL, Campbell AH, Hanten WP, Gleeson PB. Effectiveness of physical therapy for patients with neck pain: an individualized approach using a clinical decision-making algorithm. Am J Phys Med Rehabil. 2003 Mar;82(3):203-18; quiz 219-21. doi: 10.1097/01.PHM.0000052700.48757.CF. PMID 12595773
- [Result] Freburger JK, Carey TS, Holmes GM. Effectiveness of physical therapy for the management of chronic spine disorders: a propensity score approach. Phys Ther. 2006 Mar;86(3):381-94. PMID 16506874
- [Result] Hinkelmann K. Designe and análisis of experiments, Volume I, Introduction to experiment designe. 2, editor. Wiley; 2008
- [Result] Bailey A R Designe of comparative experiments. Cambridge University Press; 2008.
- [Result] Elliott SA, Brown JS. What are we doing to waiting list controls? Behav Res Ther. 2002 Sep;40(9):1047-52. doi: 10.1016/s0005-7967(01)00082-1. PMID 12296489
- [Result] Angst F, Schwyzer HK, Aeschlimann A, Simmen BR, Goldhahn J. Measures of adult shoulder function: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) and its short version (QuickDASH), Shoulder Pain and Disability Index (SPADI), American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form, Constant (Murley) Score (CS), Simple Shoulder Test (SST), Oxford Shoulder Score (OSS), Shoulder Disability Questionnaire (SDQ), and Western Ontario Shoulder Instability Index (WOSI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S174-88. doi: 10.1002/acr.20630. No abstract available. PMID 22588743
- [Result] Moshe S, Izhaki R, Chodick G, Segal N, Yagev Y, Finestone AS, Juven Y. Predictors of return to work with upper limb disorders. Occup Med (Lond). 2015 Oct;65(7):564-9. doi: 10.1093/occmed/kqv100. Epub 2015 Jul 20. PMID 26195341
- See also: DASH Outcome Measure Institute for Work & Health — http://dash.iwh.on.ca/about-dash